CLINICAL TRIAL: NCT02119845
Title: A Prospective Clinical Evaluation of the TVA FLEX-1 Device Protocol FLEX-1-001
Brief Title: A Prospective Clinical Evaluation of the Total Vascular Access (TVA) FLEX-1 Device Protocol FLEX-1-001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLEX-1-001
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Disease (CKD)
Keywords: Chronic kidney disease; Arteriovenous fistula (AVF); Hemodialysis; Vascular access; Endovascular AVF (EndoAVF)
MeSH Terms: conditions — Renal Insufficiency, Chronic; Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endovascular AVF (EndoAVF) (Experimental): The FLEX System will be used to endovascularly create a fistula in CKD patients who require hemodialysis vascular access.
  Interventions: Device: Endovascular AVF (EndoAVF)

INTERVENTIONS:
Device: Endovascular AVF (EndoAVF) — The FLEX System will be used to endovascularly create a fistula in CKD patients who require hemodialysis vascular access.
  Other Names: FLEX

SUMMARY:
The primary objective of this clinical study is to evaluate the preliminary safety and effectiveness of using the FLEX-1 device for the creation of an arteriovenous fistula (AVF) in patients requiring chronic hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for a native surgical arteriovenous fistula, as determined by the treating physician.
* Adult (age >18 years old).
* Advanced chronic kidney disease (CKD), stage 4 or 5 electing for hemodialysis.
* Written informed consent obtained

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 6 months
  The safety of the FLEX-1 system based on the overall complication rates derived from adverse event data.

SECONDARY OUTCOMES:
Access Functionality | 6 Months
  The functionality of the AVF will be measured based on use of the AVF with two needles for at least 75% of dialysis sessions over a 4-week period following at least a one month maturation period.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Ebner, MD, Principal Investigator — Italian Hospital
Locations (1):
- Italian Hospital, Asunción, Paraguay